CLINICAL TRIAL: NCT01588119
Title: Prospective Register Study to Record Safety and Efficacy of New Oral Anticoagulants
Brief Title: Register for New Oral Anticoagulants
Acronym: NOAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: NOAC
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Anticoagulation Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Dabigatran: in atrial fibrillation
- Rivaroxaban: in atrial fibrillation and VTE
- Apixaban: in atrial fibrillation and VTE
- Edoxaban: in atrial fibrillation and VTE

SUMMARY:
Patients, who are adjusted to a new oral anticoagulant (Dabigatran, Rivaroxaban, Apixaban, Edoxaban) in routine treatment will recorded in this register. Within this register a characterization of patients (with regard to demography and indication) and therapy (with regard to medication, dose and duration) will be done. On basis of defined clinical relevant end points the long-term efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* indication for treatment with long term anticoagulation
* initial adjustment or change to nex oral anticoagulant within routine treatment
* indication for treatment with long term anticoagulation within the register:
* permanent anticoagulation in arterial fibrillation
* intended anticoagulation in acute venous thromboembolism for min. 3 months
* other anticoagulation for min. 3 months within the approved indication

Exclusion Criteria:

* missing Informed Consent Form
* missing phone number for telephone follow up
* contraindication for therapy with new oral anticoagulant (Dabigatran, Rivaroxaban, Apixaban, Edoxaban) according to Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in clinical routine
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-11; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Beyer-Westendorf, MD, Principal Investigator — study site at Universitätsklinikum Dresden on behalf of GWT-TUD GmbH
Locations (1):
- Universitätsklinikum Dresden on behalf of GWT-TUD GmbH, Dresden, Germany

REFERENCES:
- [Derived] Beyer-Westendorf J, Marten S, Naue C, Tittl L, Hansel U, Beyer-Westendorf I, Mizera H, Schreier T, Festerling E, Reitter A, Spindler M, Bornhauser M. Rates, management and outcome of bleeding complications during edoxaban therapy in daily care - results from the DRESDEN NOAC REGISTRY. Thromb Res. 2020 Jun;190:91-98. doi: 10.1016/j.thromres.2020.03.021. Epub 2020 Apr 19. PMID 32335423
- [Derived] Beyer-Westendorf J, Ebertz F, Forster K, Gelbricht V, Michalski F, Kohler C, Werth S, Endig H, Pannach S, Tittl L, Sahin K, Daschkow K, Weiss N. Effectiveness and safety of dabigatran therapy in daily-care patients with atrial fibrillation. Results from the Dresden NOAC Registry. Thromb Haemost. 2015 Jun;113(6):1247-57. doi: 10.1160/TH14-11-0954. Epub 2015 Mar 5. PMID 25739533
- [Derived] Beyer-Westendorf J, Forster K, Pannach S, Ebertz F, Gelbricht V, Thieme C, Michalski F, Kohler C, Werth S, Sahin K, Tittl L, Hansel U, Weiss N. Rates, management, and outcome of rivaroxaban bleeding in daily care: results from the Dresden NOAC registry. Blood. 2014 Aug 7;124(6):955-62. doi: 10.1182/blood-2014-03-563577. Epub 2014 May 23. PMID 24859362